CLINICAL TRIAL: NCT06948474
Title: Clinical Study on the Effect of Traditional Chinese Medicine Formula Dachengqi Decoction on Early Gastrointestinal Function Recovery After Whipple Surgery
Brief Title: Dachengqi Decoction for Enhancing Early Gastrointestinal Recovery After Whipple Surgery
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Zhiying Yang, Director, Head of Hepatobiliary and Pancreatic Surgery, Clinical Professor, China-Japan Friendship Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-KY-379-1
Record Dates: First submitted 2025-03-24; First posted 2025-04-29 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Whipple Operation
Keywords: Pancreatic Cancer; IPMN, Pancreatic; whipple; Pancreaticoduodenectomy; Periampullary
MeSH Terms: conditions — Pancreatic Neoplasms; Pancreatic Intraductal Neoplasms | interventions — dachengqi decoction; Saline Solution

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dachengqi Decoction Experimental Group (Experimental): All study participants underwent intraoperative placement of modified gastrointestinal dual-lumen feeding tubes with distal ends positioned 15-20 cm distal to the gastrojejunostomy anastomosis (all devices were uniformly procured by China-Japan Friendship Hospital). Participants received Dachengqi decoction (50 ml BID) via pump infusion at 10 ml/h starting 12 hours postoperatively, continuing through postoperative days 1-3.
  Interventions: Drug: Dachengqi decoction; Procedure: modified gastrointestinal dual-lumen feeding tube
- control group (Placebo Comparator): All participants received intraoperative placement of modified gastrointestinal dual-lumen feeding tubes (15-20 cm distal to gastrojejunostomy anastomosis; devices uniformly procured by China-Japan Friendship Hospital). Participants were administered glucose and sodium chloride injection (50 ml BID) via pump infusion at 10 ml/h starting 12 hours postoperatively, continuing through postoperative days 1-3.
  Interventions: Procedure: modified gastrointestinal dual-lumen feeding tube; Drug: Normal Saline (0.9% NaCl)
- Blank control group (No Intervention): No specific therapeutic intervention was indicated

INTERVENTIONS:
Drug: Dachengqi decoction — experimental Participants received Dachengqi decoction (50 ml BID) via pump infusion at 10 ml/h starting 12 hours postoperatively, continuing through postoperative days 1-3.
  Arms: Dachengqi Decoction Experimental Group
Procedure: modified gastrointestinal dual-lumen feeding tube — experimental and control group participants underwent intraoperative placement of modified gastrointestinal dual-lumen feeding tubes with distal ends positioned 15-20 cm distal to the gastrojejunostomy anastomosis (all devices were uniformly procured by China-Japan Friendship Hospital).
  Arms: Dachengqi Decoction Experimental Group; control group
Drug: Normal Saline (0.9% NaCl) — control group participants were administered glucose and sodium chloride injection (50 ml BID) via pump infusion at 10 ml/h starting 12 hours postoperatively, continuing through postoperative days 1-3.
  Arms: control group

SUMMARY:
To investigate the clinical efficacy of the traditional Chinese medicine formula Dachengqi Decoction in promoting early gastrointestinal function recovery after Whipple surgery, and to evaluate its impact on postoperative nutritional status, hospitalization duration, and complication rates, thereby providing evidence for optimizing postoperative rehabilitation strategies in pancreaticoduodenectomy patients.

DETAILED DESCRIPTION:
Study Design: This prospective, open-label, randomized controlled trial will enroll 45 patients undergoing pancreaticoduodenectomy (PD) or pylorus-preserving pancreaticoduodenectomy (PPPD) at the study center. Participants will be divided into three groups: the experimental group (15 patients receiving Dachengqi Decoction), the control group (15 patients receiving glucose-sodium chloride solution), and a retrospective blank control group (15 historical cases). Simple randomization will be applied for group allocation.

Intervention:

Experimental Group: Dachengqi Decoction (composed of Houpu 24g, Zhishi 12g, Dahuang 12g, and Mangxiao 9g) will be prepared by the hospital pharmacy. Administered at 50 mL twice daily via jejunal tube infusion (10 mL/h), starting 12 hours postoperatively for three consecutive days.

Control Group: Glucose-sodium chloride solution (250 mL: glucose 12.5g and sodium chloride 2.25g) will be administered using the same protocol.

Blank Control Group: No additional intervention; data will be retrospectively collected from eligible historical cases.

Key Procedures:

Baseline Assessments: Preoperative evaluations include medical history, physical examinations (e.g., bowel sounds), laboratory tests (blood counts, biochemistry, coagulation, inflammatory markers), imaging (CT/MRI), and validated scales (nutritional status, mental health, gastrointestinal function).

Intraoperative Management: Standardized anesthesia and placement of a dual-lumen feeding tube distal to the gastrojejunal anastomosis.

Postoperative Monitoring: Record time to first defecation, flatus, oral intake, ambulation, vomiting frequency, bowel sounds, pain scores, and complications (e.g., delayed gastric emptying [DGE]). Imaging (abdominal CT) and laboratory tests will be performed on postoperative days 1, 3, 5, 7, and 30.

Follow-Up: Assessments at 30 days post-surgery will include gastrointestinal function, nutritional status, and adverse events.

Endpoints:

Primary Endpoints: Gastrointestinal function (evaluated via standardized scales) and nutritional status (PG-SGA score) at 1 month postoperatively.

Secondary Endpoints: Total hospitalization duration, time to gastrointestinal recovery (flatus, defecation, oral intake), and incidence of complications (e.g., DGE graded by ISGPS criteria).

Statistical Analysis: Continuous variables will be analyzed using ANOVA or non-parametric tests, while categorical variables will be assessed with chi-square or Fisher's exact tests. Linear/logistic regression and Cox models will be applied for outcome analysis. A sample size of 15 per group was calculated (power=0.9, α=0.05).

Ethics and Compliance: The study protocol and informed consent forms will be approved by the institutional ethics committee. Participants or their legal representatives must provide written consent. Confidentiality of patient data will be maintained, and results will be disseminated through peer-reviewed publications.

Timeline: Patient enrollment is scheduled for completion by March 1, 2026, with final results expected by June 1, 2026.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-75 years, regardless of gender (n=45);
* Meeting American Society of Anesthesiologists (ASA) physical status classification I-II criteria, scheduled to undergo pancreaticoduodenectomy or pylorus-preserving pancreaticoduodenectomy under combined intravenous-inhalational general anesthesia;
* No participation in other clinical trials within 6 months prior to the study initiation;
* Absence of severe preexisting cardiac, neurological, renal, endocrine, or hematologic diseases that may affect surgical outcomes or postoperative prognosis (e.g., unstable angina, heart failure, uncontrolled hypertension, severe neuropathy, psychiatric disorders, renal insufficiency, diabetes, hematologic disorders, severe alcoholic liver disease, substance abuse, or alcoholism);
* Participants free of cognitive impairment, aphasia, or psychiatric disorders, possessing intact communication skills and capable of comprehending and signing the informed consent form.

Exclusion Criteria:

* Patients aged <18 or >75 years;
* Not meeting American Society of Anesthesiologists (ASA) physical status classification I-II criteria;
* History of severe cardiac, neurological, renal, endocrine, or hematopoietic comorbidities that may impact surgical outcomes or postoperative prognosis (e.g., unstable angina, heart failure, uncontrolled hypertension, severe neuropathy, psychiatric disorders, renal insufficiency, diabetes, hematologic diseases, severe alcoholic liver disease, substance abuse, or alcoholism);
* Participants in either treatment group refusing to sign informed consent forms;
* Participation in other clinical trials within 6 months prior to study initiation;
* Patients deemed by investigators unsuitable for efficacy evaluation or unlikely to complete treatment course and follow-up.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
One month postoperative evaluation of gastrointestinal function | 1 month after surgery
  assessed through three independent systems: Functional bowel recovery: Evaluated through I-FEED scoring system (0-10; lower score reflects better postoperative recovery)

SECONDARY OUTCOMES:
postoperative assessment of gastrointestinal functional recovery | From surgery date through postoperative day 30.
  Time to first flatus (hours) Time to first bowel movement (hours) Time to oral intake initiation (hours) Time to first ambulation (hours)

CONTACTS AND LOCATIONS:
Locations (1):
- China-Japan Friendship Hospital, Beijing, Beijing Municipality, China